CLINICAL TRIAL: NCT02154971
Title: Assessment of Age-related Hearing Loss in HIV-1 Patients
Acronym: HELO
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: AMR_2013-10
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: HIV Seropositivity
Keywords: HIV Seropositivity; Audiometry; Hearing Loss
MeSH Terms: conditions — HIV Seropositivity; Hearing Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: HIV infected for more than 10 years, aged over 40, treated with antiretroviral therapy
- Control: non-HIV (matched for age and gender)

SUMMARY:
The ageing process is known to be accelerated in HIV-infected patients, compared to the general population.

Normal age-related hearing loss (presbyacusia) is a frequent phenomenon, affecting more than 70% of people above 65 years. It is believed to be mostly the consequence of a mitochondrial damage caused by oxidative stress.

Risk factors for accelerated age-related hearing loss are present in many HIV-infected patients : chronic inflammation, smoking, diabetes, etc.

The global aim is to measure the prevalence of presbyacusia in a well controlled HIV positive population in France, and to compare it to HIV negative controls matched for age and sex.

90 HIV positive patients and 90 age- and sex- matched HIV negative controls will undergo a screening for presbyacusia (pure-tone, speech and evoked-response audiometry).

We expect to find an increased prevalence of presbyacusia in HIV-infected patients, as compared to controls matched for age and sex.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years and more
* HIV-1 infection known since 10 years and more
* Undetectable plasmatic HIV-1 viral load thanks to antiretroviral therapy (any regimen) for at least 5 years
* CD4 lymphocytes count above 350
* Condition of Cerebral Small Vessel Disease detected recently with MRI

Exclusion Criteria:

* Personal history of otologic pathology or otologic surgery
* Family history of hearing impairment
* Personal history of bacterial meningitis
* Personal history of neurological disease
* Personal history of treatment with ototoxic drugs
* Personal history of treatment with chemotherapy
* Use of illegal drugs (except cannabis or poppers)
* Alcoholism
* Diabetes complicated by retinopathy and/or by glomerular filtration rate < 60 mL/min and/or by proteinuria > 300 mg)
* Uncontrolled high blood pressure (WHO criteria)
* MRI contraindication
* Known pregnancy or breastfeeding woman
* No medical insurance coverage

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed for HIV infection in the department of infectious diseases of Saint-Antoine hospital or Bichat hospital and/or by a private HIV-specialized physician in Paris, France
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2013-11-18 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
hearing loss at several frequencies | Baseline
  Measurement by audiometry (pure tone and speech audiometry at 500Hz, 1000Hz, 2000Hz, 3000Hz and 8000 Hz), expressed in dB.

SECONDARY OUTCOMES:
threshold for speech intelligibility | Baseline
  measured by speech audiometry
Proportion of patients with neuropathic hearing loss | Baseline
Interval I-V on the evoked-response audiogram | Baseline
Maximum speech intelligibility | Baseline
  Measured by speech audiometry
Proportion of patients with age-related hearing loss | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Moulignier, MD, Principal Investigator — Fondation Ophtalmologique Antoine de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, Île-de-France Region, France